CLINICAL TRIAL: NCT06921954
Title: Study Effects of the PRECAPP System on Precarious and Vulnerable Pregnant Women
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0087_MATER_PRECAPP
Record Dates: First submitted 2025-02-27; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pregnant Women; Vulnerable Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (3):
- 1st stage: preliminary study 4 to 5 PRECAPP files: Construction of an analysis grid including :
  * Patient characteristics (age, nationality, number of children, family situation, etc.)
  * Number of months pregnant at the time of inclusion in PRECAPP
  * Reasons for referral and inclusion in the program
  * Characterization of vulnerability and precariousness
  * Nature of care: what follow-up is in place? (Distinction between "classic" follow-up and PRECAPP-specific follow-up)
  * What problems have been anticipated and are likely to have been avoided during pregnancy, childbirth and after childbirth?
  * What difficulties have been encountered that have not been fully or partially overcome?
  Study of 4 to 5 files selected by the PRECAPP team, representing "typical" PRECAPP situations in 2023.
  This stage will enable us to establish an initial typology and target the files to be studied in subsequent stages.
- 2nd stage: in-depth analysis of 15 to 20 PRECAPP files: * Random selection of files in each PRECAPP category ("classic follow-up" files and "late follow-up" files)
  * Data collection from files
  * The analysis grid will serve as a framework for in-depth examination of the files. It may, of course, be fine-tuned along the way, in line with the qualitative nature of the research-intervention approach.
- Step 3: Analysis of 4 to 5 maternity files (not monitored by PRECAPP): Selection of 4-5 files of precarious and vulnerable women who were not monitored by PRECAPP and who arrived at the maternity hospital without PRECAPP's intervention, in collaboration with the maternity hospital and PRECAPP.
  Construction of a specific analysis grid (different from the analysis grid for PRECAPP files, including in particular the reasons why patients escaped PRECAPP follow-up).
  Data collection and in-depth analysis of files (maternity unit and research team)

SUMMARY:
The themes of city-hospital coordination, patient pathways and the decompartmentalization of the city-hospital-medical-social and social sectors are becoming a major preoccupation for the healthcare sector, and a key factor in its dynamic transformation. A number of initiatives taken in this direction, either by the regulatory authorities (development of tools to promote coordination between healthcare professionals), by hospital establishments or by city professionals (notably CPTS), attest to a growing interest in the subject.

The École des Mines de Paris, whose highly collaborative research methods (research-intervention) are anchored in concrete support for transformation projects, and the University of Lille (LUMEN) are thus increasingly called upon to support players in these areas.

In this context, collaborative work with a Quebec research team (Ecole Nationale d'Administration Publique and Université de Sherbrooke) was launched in 2023 to compare forms of healthcare pathway management between two different healthcare systems, and their effects on vulnerable people (elderly, disabled, migrants, homeless, etc.). In France, the quantitative component is based on the use of PMSI databases, and aims to analyze the characteristics of "abnormally long" patient stays, in order to identify variables (relating either to patients or to care) likely to explain longer lengths of stay. The qualitative component is based on interviews with professionals and the reconstruction of patient pathways marked by breaks in care. The aim is to understand the very notion of breakdowns, the mechanisms by which they occur and the strategies put in place to avoid or deal with them.

Collaboration with the PRECAPP research team

As part of the qualitative component of the research program, the French team met several times between February and summer 2024 with members of the PRECAPP program. The PRECAPP system's function (to support vulnerable pregnant women in the perinatal period) and its mission (to identify the risks of disruption to care as early as possible in pregnancy, and to coordinate care during pregnancy and in the postnatal period) are at the heart of the Franco-Quebec research.

An initial working meeting between the PRECAPP team and the researchers provided an opportunity to describe the system and to demonstrate that its operation and the specific support it provides make it possible to anticipate certain difficulties in the care of women (before, during and after birth) and to help avoid disruptions in care.

The PRECAPP system is therefore fully in line with a comprehensive approach to the perinatal care of precarious and vulnerable women. This care concerns intra-hospital care, but it also contributes to the decompartmentalization of city-hospital care.

It is with the aim of highlighting the contributions of the PRECAPP system to the quality of care provided, the limits to its action, and to assess the way in which it helps to avoid breakdowns, that a collaboration between researchers and practitioners has been set up and will enable this study to be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Follow-up in 2023 at Gonesse Hospital
* Patient having started her PRECAPP follow-up in 2023, between the 2nd and 5th month of pregnancy and having been accompanied throughout her PRECAPP journey (before, during and after childbirth): Classic" PRECAPP pathway
* Patient with integration (in 2023) of the PRECAPP program late in pregnancy (up to 1 month before delivery): PRECAPP "late" pathway
* Vulnerable and precarious patient not followed by PRECAPP but who should have been (maternity course completed in 2023): PRECAPP "non-integration" pathway

Exclusion Criteria:

* Patient without vulnerability/poverty
* Patient not followed at the CHG in 2023

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age ≥ 18 years
  * Follow-up in 2023 at Gonesse Hospital
  * Patient having started her PRECAPP follow-up in 2023, between the 2nd and 5th month of pregnancy and having been accompanied throughout her PRECAPP journey (before, during and after childbirth): Classic" PRECAPP pathway
  * Patient with integration (in 2023) of the PRECAPP program late in pregnancy (up to 1 month before delivery): PRECAPP "late" pathway
  * Vulnerable and precarious patient not followed by PRECAPP but who should have been (maternity course completed in 2023): PRECAPP "non-integration" pathway
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
demographics | enrollment
  age, nationality, number of children, family situation
clinics | enrollment
  stage of pregnancy, reason for referral, characterization of vulnerability and precariousness, problems anticipated and avoided, difficulties encountered and overcome

SECONDARY OUTCOMES:
follow up | enrollment
  Nature of support